## **Written Informed Consent**

## Safety and Suitability of ICL for Correction of Refractive Errors Without the Use of Dispersive OVDs

Priciple investigator Sohaib Ahmed Mahmood, MD

Practicing ophthalmologist

Ibn Al-Haithem teaching eye hospital

Author Sohaib Ahmed Mahmood, MD

Practicing ophthalmologist

Ibn Al-Haithem teaching eye hospital

NCT identifier NCT06371079

Unique protocol ID NO-OVD-ICL

Date 12-21-2021

## Informed Consent for Cataract Surgery and Intraocular Lens Implantation

## **Authorization and Consent for Surgery**

I, the undersigned, ......, hereby authorize Dr. Sohaib Ahmed to perform cataract surgery and implant an intraocular lens.

I have understood all the necessary information about my treatment and that the doctor has answered all my questions about the treatment in a clear and satisfactory manner. I have received a copy of this document.

I have decided of my own free will to consent to this surgical procedure and any other procedure that the doctor deems appropriate during the surgery. I specifically acknowledge that I have understood and accepted the following:

- Possible complications ranging from mild eye inflammation to severe vision loss or impairment.
- I am fully aware of the risks that may arise from or during the operation and I bear full responsibility in this regard.
- I agree and clearly agree that the surgeon and the hospital do not bear any responsibility for the failure of the operation.
- The hospital and the doctor do not guarantee the success of the operation in any way.
- I am aware that the hospital has provided the surgeon with the latest medical equipment to perform the operation.
- Corneal swelling (or edema) may occur: This swelling is usually caused by the implanted lens or by the insertion of surgical instruments into the eye. It may appear a few hours after the operation and vision may become blurred somewhat due to this corneal swelling. It usually disappears on its own or may require corneal replacement.
- Increased eye pressure: Eye pressure may increase slightly after surgery because some of the fluids used during surgery do not pass through the natural drainage channels of the eye as expected. This condition usually manifests as a headache or severe pain in the eye area. Intraocular pressure-lowering medications may be prescribed during the postoperative period. In any case, the eye drops prescribed by the doctor will help to alleviate these complications and may require cataract surgery.
  - Bleeding: This is a very rare possibility but can still occur.

- Retinal detachment may occur: People with severe myopia are more prone to retinal detachment than others.
- Infection may occur, although the use of antibiotic eye drops makes the possibility of infection very low.
- The patient needs to follow up regularly as the doctor sees fit and any noncompliance with regular follow-up may lead to serious complications.
  - The doctor may need to replace or modify the lens.
- Dryness may occur and most cases are resolved with artificial tears or, in rare cases, surgery to reduce dryness.
- The goal of the operation is to replace or reduce glasses as much as possible, i.e. in rare cases the patient may need glasses to improve vision for distant objects or reading glasses or both.

| Patient's Name and Signature: |
|-------------------------------|
| Date |
| Witness: |
| Date |